CLINICAL TRIAL: NCT01856855
Title: RAD 1203: Pilot Trial Evaluating Stereotactic Body Radiotherapy With Integrated Boost for Clinically Localized Prostate Cancer
Brief Title: Pilot Trial Evaluating Stereotactic Body Radiotherapy With Integrated Boost for Clinically Localized Prostate Cancer (RAD 1203)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Fiveash, MD (Other)
Responsible Party: Sponsor-Investigator, John Fiveash, MD, Professor and Vice Chair, University of Alabama at Birmingham Department of Radiation Oncology, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F121218006
Record Dates: First submitted 2013-04-10; First posted 2013-05-17 (Estimated); Results first posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Radiation Toxicity; Sexual Dysfunction
Keywords: Prostate Cancer; Prostate Adenocarcinoma; Radiation; SBRT; Stereotactic Body Radiation Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries; Sexual Dysfunction, Physiological | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Body Radiation Therapy with Integrated Boost (Experimental)
  Interventions: Radiation: Stereotactic Body Radiation Therapy with Integrated Boost

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy with Integrated Boost — SBRT with Integrated boost at 7.25 Gy and 8.00 Gy per fraction for five fractions
  Other Names: SBRT; IMRT; VMAT

SUMMARY:
This study will investigate the safety, tolerability, and effectiveness of giving a higher dose to the part of the prostate which contains the cancer while giving a standard radiation dose to the entire prostate. The investigators have hypothesized that this treatment technique will effectively control the prostate cancer while minimizing the side effects.

DETAILED DESCRIPTION:
Objectives:

Primary

-Clinically assess the early toxicity of SBRT with integrated boost for clinically localized prostate cancer

Secondary

* Determine the technical feasibility of stereotactic body radiotherapy (SBRT) with integrated boost for clinically localized prostate cancer

  * Determine the treatment planning and dosimetric feasibility
  * Evaluate the treatment delivery quality assurance
* Clinically assess early efficacy, late toxicity, and quality of life for patients receiving SBRT with integrated boost for clinically localized prostate cancer

Patients will undergo 5 total radiation treatments over 7-17 day period.

Patients will be asked to complete American Urological Association Symptom Index (AUA SI), Sexual Health Inventory of Men (SHIM), and the Expanded Prostate Index Composite (EPIC)questionnaires. The EPIC assesses bowel, urinary, and sexual function. These questionnaires will be completed at the following time points: Baseline, AUA SI will be collected on the last day of treatment, and every 3 months for the first year following the start of radiation, then every 6 months for year 2.

After completion of study therapy, patients are followed-up every 3 months for the first year, then every 6 months for year 2.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have Histologically confirmed prostate adenocarcinoma, with biopsies obtained within twelve months of patient registration
* NCCN risk category very low, low, or intermediate risk
* Combined Gleason score <7
* PSA within three months of enrollment < 20ng/ml
* Clinical stage T1a-c N0M0 or clinical stage T2aN0M0
* Life expectancy > 5 years
* Risk of malignant lymph node involvement < 15% as calculated on Partin tables
* Karnofsky performance status (KPS) > 60
* Age > 19 years
* Subjects given written informed consent

Exclusion Criteria:

* History of inflammatory bowel disease
* Prior radical prostate surgery, transurethral resection of the prostate(TURP), or prostate cryotherapy
* Patients using immunosuppressive medications or other medications that may increase radiation toxicity such as methotrexate, sirolimus, tacrolimus, or colchicine that are unable to discontinue these medications during SBRT course. Use of corticosteroids are not considered an exclusion criteria.
* Platelet count < 70
* Patients unable to discontinue anti-platelet or anti-coagulant medicine such as clopidogrel, dabigatran, warfarin, or low molecular weight heparin. Use of aspirin is not an exclusion criteria.
* Pre-SBRT prostate volume > 120 cc as estimated by trans-rectal ultrasound at time of prostate biopsy (TRUS biopsy).
* Risk of malignant lymph node involvement > 15% as calculated on Partin tables.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-02; Primary Completion 2021-12 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John B Fiveash, MD, Principal Investigator — University of Alabama at Birmingham Radiation Oncology
Locations (1):
- Hazelrig-Salter Radiation Oncology Center, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stereotactic Body Radiation Therapy With Integrated Boost
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Body Radiation Therapy With Integrated Boost
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced Early Toxicity of SBRT With Integrated Boost for Localized Prostate Cancer
Description: Early toxicity (defined as events occurring within 90 days of therapy) will be assessed by physician history and physical exams and patient toxicity/quality-of-life questionnaires to be administered at regular intervals.
Time Frame: Within 3 months of the completion of radiation therapy
Measure: Number; unit: number of participants
Arm/Group | Stereotactic Body Radiation Therapy With Integrated Boost
Number analyzed (Participants) | 26
number of participants | 22

2. Secondary Outcome: Treatment Planning Feasibility
Description: Feasibility will be defined as the ability of the treatment planner to create a plan that meets the following criteria:
  * 100% of radiation target prescription (36.25 Gy) covers greater than or equal to 95% of the target (prostate)
  * At least 95% of the boost prostate (area within the prostate most likely harboring cancer) prescription (38.0 Gy) covers 95% of this boost target volume
  * All normal tissue dose constraints are met -i.e., nearby rectum, bladder, and femoral heads do not exceed the recommended radiation dose limits
  If the physician must utilize a plan that compromises target coverage or normal tissue dose constraints to levels not meeting the criteria above, then the plan will be scored as not meeting technical feasibility requirements.
Time Frame: Within 6 months of completion of radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiation Therapy With Integrated Boost
Number analyzed (Participants) | 26
Participants | 26

3. Secondary Outcome: Early Efficacy
Description: Efficacy will be defined as the absence of biochemically detected (via PSA lab testing) prostate cancer or clinically detected prostate cancer at each interval follow-up visit (every three months for year one, then every 6 months for year two after treatment). "Absence of prostate cancer" is defined as no evidence of tumor recurrence by two methods:
  1. No prostate cancer recurrence evident on the physical examination performed by the physician.
  2. No rise in the PSA more than 2 ng/ml above the lowest PSA value ever obtained pre or post treatment. A rise in the PSA more than 2 ng/ml from a patient's lowest value is the standard definition for post-radiation PSA biochemical prostate cancer failure.
Time Frame: Within 6 months of completion of radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiation Therapy With Integrated Boost
Number analyzed (Participants) | 26
Participants | 26

4. Secondary Outcome: Number of Patients Who Experienced Late Toxicity
Description: Late toxicity (defined as toxicity occuring >90 days after treatment) will be assessed with regular clinical exams and patient toxicity questionnaires.
Time Frame: Within 6 months of completion of radiation therapy
Measure: Number; unit: number of participants
Arm/Group | Stereotactic Body Radiation Therapy With Integrated Boost
Number analyzed (Participants) | 26
number of participants | 22

5. Secondary Outcome: Median Quality of Life Score
Description: Median of quality of life score will be assessed with regular clinical exams and patient quality of life questionnaires (American Urologic Association Symptom Index score ranges from 0 to 35 with the higher scores indicating more severe, Sexual Health Inventory score ranges from 1 to 25 with 1 being severe and 25 being no signs, Extended Prostate Cancer Index Composite- Bowel, Extended Prostate Cancer Index Composite- Urinary, and Extended Prostate Cancer Index Composite- Sexual scales range from 1 (worst) to 100 (best)).
Time Frame: Within 6 months of completion of radiation therapy
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Stereotactic Body Radiation Therapy With Integrated Boost
Number analyzed (Participants) | 26
score on a scale
  American Urologic Association Symptom Index | 11 [0 to 35]
  Sexual Health Inventory for Men | 17 [1 to 25]
  Extended Prostate Cancer Index Composite-Urinary | 85.8 [1 to 100]
  Extended Prostate Cancer Index Composite-Sexual | 57.7 [1 to 100]
  Extended Prostate Cancer Index Composite-Bowel | 91.1 [1 to 100]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Stereotactic Body Radiation Therapy With Integrated Boost
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 22/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Body Radiation Therapy With Integrated Boost (N=26)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Hematochezia (Gastrointestinal disorders) | 3 (3)
Dysuria (Renal and urinary disorders) | 7 (7)
Urinary Retention (Renal and urinary disorders) | 2 (2)
Urinary Urgency (Renal and urinary disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT01856855/Prot_SAP_000.pdf